CLINICAL TRIAL: NCT00113737
Title: Fluoxetine as a Quit Smoking AID for Depression Prone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Masking: Double | Purpose: Prevention
Other Study IDs: 183; R01HL059348 (NIH)
Record Dates: First submitted 2005-06-09; First posted 2005-06-10 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2005-06

CONDITIONS: Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases | interventions — Fluoxetine; Cognitive Behavioral Therapy

INTERVENTIONS:
Drug: fluoxetine
Behavioral: cognitive behavioral therapy

SUMMARY:
To test whether adding fluoxetine pharmacotherapy to behavioral cessation treatment improves the depression-prone smoker's ability to quit.

DETAILED DESCRIPTION:
DESIGN NARRATIVE:

The research was a treatment-matching study to test whether adding fluoxetine pharmacotherapy to behavioral cessation treatment improved the depression-prone smoker's ability to quit. The investigators randomized 144 smokers with a prior history of depression and 206 smokers who lack such a history to a double-blind treatment with either 60 mg fluoxetine or placebo, while they underwent cognitive behavioral treatment to quit smoking. The main study outcome was biologically verified abstinence 6 months after treatment. The administration of placebo and fluoxetine began 3 weeks before the quit smoke date and continued for 2 months post-quit date (totaling 11 weeks on drug/placebo). Cognitive behavioral treatment were weekly before quitting and biweekly after quitting. There were monthly follow-up evaluations for six months after the quit date. The research tested both the Selective Benefit Hypothesis and the Generalized Benefit Hypothesis of fluoxetine's effects. The hypothesis of the mechanism of action was that the drug diminished compulsive smoking behavior, obsessional cigarette craving, and nicotine withdrawal dysphoria that occurred independently of depressive vulnerability.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
An estimated 144 smokers with a prior history of depression and 206 smokers who lacked such a history.

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1998-02; Study Completion 2002-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie Spring — U.S. Dept/Vets Affairs Med Ctr.

REFERENCES:
- [Background] Hitsman B, Spring B, Wolf W, Pingitore R, Crayton JW, Hedeker D. Effects of acute tryptophan depletion on negative symptoms and smoking topography in nicotine-dependent schizophrenics and nonpsychiatric controls. Neuropsychopharmacology. 2005 Mar;30(3):640-8. doi: 10.1038/sj.npp.1300651. PMID 15647750
- [Background] Sanchez-Johnsen LA, Fitzgibbon ML, Ahluwalia JS, Spring BJ. Eating pathology among Black and White smokers. Eat Behav. 2005 Feb;6(2):127-36. doi: 10.1016/j.eatbeh.2004.08.011. PMID 15598599
- [Background] Holmes EW, Russell PM, Kinzler GJ, Reckard CR, Flanigan RC, Thompson KD, Bermes EW Jr. Oxidative tryptophan metabolism in renal allograft recipients: increased kynurenine synthesis is associated with inflammation and OKT3 therapy. Cytokine. 1992 May;4(3):205-13. doi: 10.1016/1043-4666(92)90057-x. PMID 1498255
- [Background] Cook JW, Spring B, McChargue DE, Borrelli B, Hitsman B, Niaura R, Keuthen NJ, Kristeller J. Influence of fluoxetine on positive and negative affect in a clinic-based smoking cessation trial. Psychopharmacology (Berl). 2004 Apr;173(1-2):153-9. doi: 10.1007/s00213-003-1711-8. Epub 2004 Jan 15. PMID 14727000
- [Background] Spring B, Pagoto S, McChargue D, Hedeker D, Werth J. Altered reward value of carbohydrate snacks for female smokers withdrawn from nicotine. Pharmacol Biochem Behav. 2003 Sep;76(2):351-60. doi: 10.1016/j.pbb.2003.08.008. PMID 14592688
- [Background] Spring B, Pingitore R, McChargue DE. Reward value of cigarette smoking for comparably heavy smoking schizophrenic, depressed, and nonpatient smokers. Am J Psychiatry. 2003 Feb;160(2):316-22. doi: 10.1176/appi.ajp.160.2.316. PMID 12562579
- [Background] Johnsen L, MacKirnan D, Spring B, Pingitore R, Sommerfeld BK. Smoking as subculture? Influence on Hispanic and non-Hispanic White women's attitudes toward smoking and obesity. Health Psychol. 2002 May;21(3):279-87. doi: 10.1037//0278-6133.21.3.279. PMID 12027034
- [Background] Hitsman B, Spring B, Borrelli B, Niaura R, Papandonatos GD. Influence of antidepressant pharmacotherapy on behavioral treatment adherence and smoking cessation outcome in a combined treatment involving fluoxetine. Exp Clin Psychopharmacol. 2001 Nov;9(4):355-62. doi: 10.1037//1064-1297.9.4.355. PMID 11764011
- [Background] Richmond M, Spring B, Sommerfeld BK, MeChargue D. Rumination and cigarette smoking: a bad combination for depressive outcomes? J Consult Clin Psychol. 2001 Oct;69(5):836-40. doi: 10.1037//0022-006x.69.5.836. PMID 11680561
- [Background] Borrelli B, Spring B, Niaura R, Kristeller J, Ockene JK, Keuthen NJ. Weight suppression and weight rebound in ex-smokers treated with fluoxetine. J Consult Clin Psychol. 1999 Feb;67(1):124-31. doi: 10.1037//0022-006x.67.1.124. PMID 10028216